CLINICAL TRIAL: NCT00315263
Title: Genomics, SNPs, and Clinical Neonatology
Brief Title: Genomics, Single Nucleotide Polymorphisms (SNPs), and Clinical Neonatology
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Collaborators: University of Kansas (Other)
Responsible Party: William Truog, MD, Principal Investigator, The Children's Mercy Hospitals and Clinics
Other Study IDs: 01.3965
Record Dates: First submitted 2006-04-14; First posted 2006-04-18 (Estimated); Last update posted 2011-08-26 (Estimated); Status verified 2011-08

CONDITIONS: Lung Disease; Brain Injury; Necrotizing Enterocolitis; Respiratory Failure
Keywords: DNA; Genomics; SNPs; Neonatology; Chronic Lung Disease; Periventricular Brain Injury; Hypoxic Respiratory Failure
MeSH Terms: conditions — Lung Diseases; Brain Injuries; Enterocolitis, Necrotizing; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This research seeks to establish a neonatal DNA Tissue Bank to find out if differences in small segments of DNA predispose babies to Chronic Lung Disease (CLD), Periventricular Brain Injury (PVI), Necrotizing Enterocolitis (NEC), or Hypoxic Respiratory Failure (HRF).

DETAILED DESCRIPTION:
This genetic predisposition study does not involve investigational drugs, devices, or treatments. Our broad goal is to identify genomic factors, which contribute to the development or exacerbation of common and critical illnesses that affect preterm and near-term infants. We seek to accomplish this goal in the following ways:

* First: to test candidate gene DNA variations and link already identified single nucleotide polymorphisms (SNPs) producing functional alterations to the risk of clinically important disorders.
* Second: to utilize a whole-genomic approach to identify SNPs not previously linked to the risk of development or progression of neonatal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Less than 34 weeks gestation and less than 1500 g at birth
* Greater than or equal to 36 weeks gestation and either with hypoxic respiratory failure or with mild respiratory distress never requiring assisted ventilation

Exclusion Criteria:

* Life threatening anomalies of any organ system (e.g., cardiac, thoracic, lethal, or non-lethal chromosomal abnormalities)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intensive Care Nursery
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William E Truog, MD, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (2):
- United States (2):
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Truman Medical Center, Kansas City, Missouri

REFERENCES:
- See also: Official Web Address of sponsoring organization — http://www.childrens-mercy.org